CLINICAL TRIAL: NCT05667103
Title: The Safety and Efficacy of Mechanical Thrombectomy Using Embotrap Stent Retriever in Treating Acute Ischemic Stroke Patients
Brief Title: The Safety and Efficacy of Embotrap in Treating Acute Ischemic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Embotrap
Record Dates: First submitted 2022-11-21; First posted 2022-12-28 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2022-11

CONDITIONS: Stroke; Acute Ischemic Stroke
Keywords: Embotrap; Acute ischemic stroke; Mechanical thrombectomy; Stent retriever
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, parallel cohort study. The patients with acute middle cerebral artery occlusion were divided into Embotrap group and control group at a ratio of 1:1 to receive mechanical thrombectomy. The patients in control group will receive thrombectomy using stent retriever without inner channel approved by FDA or NMPA. Several aspects such as first-pass recanalization rate, the successful recanalization rate, and mRS score at 90 days will be compared between the two groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embotrap stent retriever (Experimental)
  Interventions: Device: Embotrap stent retriever
- Other stent retriever without endochannel (Active Comparator)
  Interventions: Device: Solitaire FR, Trevo stent retriever without inner channel

INTERVENTIONS:
Device: Embotrap stent retriever — Embotrap has a novel design of an open outer cage for clot capture and a closed inner channel for clot stabilization, with great thrombus fixation and anti-escape ability, to improve the successful recanalization rate and good prognosis of patients.
  Arms: Embotrap stent retriever
Device: Solitaire FR, Trevo stent retriever without inner channel — Other stent retriever without inner channel, such as Solitaire FR, Trevo, and other stent retrievers approved by FDA or NMPA.
  Arms: Other stent retriever without endochannel

SUMMARY:
This is a prospective, multicenter, cohort study aiming to compare the safety and efficacy of Embotrap stent retriever to other stent retrievers without inner channel for acute middle cerebral artery occlusion (MCAO). All enrolled patients will be followed up at 90 days after randomization.

DETAILED DESCRIPTION:
AIS due to large vessel occlusion (LVO) remains a substantial cause of mortality and morbidity. Recent guidelines have recommended MT as the first-line therapy for AIS-LVO in the anterior circulation. Thrombectomy using a stent retriever is safe and effective in the treatment of AIS. As a new generation of stent retriever, Embotrap stent retriever has a unique design including an open outer cage for clot capture and a closed inner channel for clot stabilization. Previous studies showed Embotrap stent retriever can achieve a successful recanalization of 88% and favorable outcome of 51%. Also, the Multicenter ARISE II Study showed the first-pass effect of EmboTrap stent retriever was 40.1%, higher than other stent retrievers, such as Solitaire FR and Trevo device. But most studies were single-armed without direct comparison. Thus, this prospective cohort study is designed to compare the safety and efficacy of Embotrap stent retriever with other stent retrievers without inner channel.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with symptoms due to acute middle cerebral artery occlusion (MCAO) treated with MT with or without intravenous thrombolysis.
2. Premorbid mRS 0-2
3. Ages 18-80 years
4. NIHSS ≥6 at admission
5. The time from onset to groin puncture ≤ 24 hours
6. ASPECTS 6-10 on non-contrast CT (NCCT) scan, MRI or CT-Perfusion (CTP)
7. Informed consent approved by patients or acceptable patient surrogate.

Exclusion Criteria:

1. Any intracranial hemorrhage or severe cerebral infarction on CT or MRI (ASPECTS < 6 points, core infarct volume ≥ 70mL or core infarct area >1/3 middle cerebral artery territory).
2. Severe allergy to contrast media allergy and nitinol
3. Refractory hypertension (SBP > 185 mmHg or DBP > 110 mmHg)
4. Platelet count < 30 x 10^9 / L
5. Coagulopathy history or hemorrhage disorders disease
6. Concurrent participation in a study involving an investigational drug or device that would impact the current study
7. Evidence of intracranial hemorrhage or hemorrhagic transformation before thrombectomy
8. Unable to complete the study and follow-up due to mental disorders, cognitive or emotional disorders
9. Pregnant or lactating women
10. Anticipated life expectancy < 6 months
11. Patients without a legally authorized representative to sign the consent form
12. For other reasons, the researchers believe that the patient is not suitable for enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
First-pass complete recanalization rate | intraoperative (After first-pass thrombectomy)
  FPE, eTICI≥2c

SECONDARY OUTCOMES:
First-pass successful recanalization rate | intraoperative (After first-pass thrombectomy)
  mFPE, eTICI≥2b50
Final successful recanalization rate | intraoperative (Final Digital Subtraction Angiography (DSA) during operation)
  mFPE, eTICI≥2b50
Final complete recanalization rate | intraoperative (Final Digital Subtraction Angiography (DSA) during operation)
  FPE, eTICI≥2c
90-day favorable outcome rate | 90-days (±14days)
  Modified Rankin scale (mRS), the scale runs from 0 to 6, running from perfect health without symptoms to death. 90-day favorable outcome is identified as mRS 0-2.
The improvement of the NIHSS scores 24 hours after surgery | 24 hours after surgery
  National Institutes of Health Stroke Scale (NIHSS)
The improvement of the NIHSS scores 5-7 days after surgery or at discharge | 5-7 days after surgery or at discharge, whichever came first
  National Institutes of Health Stroke Scale (NIHSS)
The rescue therapy rate | During procedure time
  The rate of rescue therapy, such as balloon dilation, stent implantation, and intra-arterial thrombolysis.
FFR after 5 minutes of mechanical thrombectomy | 5 minutes after successful vessel recanalization.
  Fractional flow reserve (FFR)

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, Dr., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University., Beijing, China